CLINICAL TRIAL: NCT06096935
Title: Exome Evaluation in Patients Living with Diabetes Complicated by Charcot Neuroarthropathy.
Acronym: CHARCOTEX
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/0025
Record Dates: First submitted 2023-10-16; First posted 2023-10-24 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes
Keywords: type 2 Diabetes; CHARCOT neuroarthropathy; Exome
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: patients with type 2 diabetes complicated by active or chronic Charcot neuropathy
  Interventions: Other: bood sample
- Group 2: patients living with type 2 diabetes without active or chronic Charcot neuroarthropathy.
  Interventions: Other: bood sample

INTERVENTIONS:
Other: bood sample — Exome measurements

SUMMARY:
Diabetes, like obesity, has reached worldwide proportions such that we're talking about a pandemic. These two diseases are a major cause of mortality and multiple complications. The medical and financial stakes involved make these two diseases a major public health issue. Two groups of factors contribute to these diseases: the environment and genetics. The use of next-generation sequencing (NGS) is a highly relevant tool for identifying mutations in already known genes, or new genes involved in the disease, for diagnostic purposes. This approach makes it possible to validate previously described genes and/or discover new loci linked to new signalling pathways involved in the pathophysiology of Charcot's foot in patients with diabetes

DETAILED DESCRIPTION:
In patients living with diabetes, a rare and devastating joint complication known as Charcot's neuroarthropathy (CN) has been observed. The clinical presentation of this complication is characterized by activation of inflammation and bone remodeling markers, disruption of the osteoblast and osteoclast system, activation of the RANKL (Receptor activator of nuclear factor-kappa B ligand) system and its antagonist osteoprotegerin (OPG), and often a fatigue fracture due to physical activity.

The pathogenic mechanisms of CN have been the subject of much debate, and there are a number of competing theories which are not necessarily exclusive.

CN patients have been shown to have reduced bone density in the lower limbs compared with neuropathic subjects. Studies using bone markers to assess bone formation and resorption demonstrated that there is an increase in osteoclastic activity relative to osteoblastic activity in both acute and chronic forms of CN. In 2007, W.J. Jeffcoate described CN as an increased inflammatory response to injury inducing increased bone lysis. Since the emergence of this theory, a significant number of studies have evaluated inflammatory factors and bone modeling in patients with CN, such as C-reactive protein, TNF α and IL6. Three studies showed an increase in their levels in the setting of CN.

otherwise known genes, or new genes implicated in the disease, for diagnostic purposes This approach makes it possible to validate previously described genes and/or discover new loci linked to new signalling pathways involved in the pathophysiology of Charcot's foot in patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 to 70
* with type 2 diabetes for at least one year
* with active or chronic Charcot neuroarthropathy (Group 1) OR
* never had Charcot neuroarthropathy (Group 2)
* Have agreed to participate in the study and have signed an informed consent form.

Exclusion Criteria:

- Subject under guardianship or curatorship.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patiens living with type 2 diabetes complicates by Charcot Neuroarthopathy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-07-11 (Actual); Primary Completion 2025-01-18 (Actual); Study Completion 2025-01-18 (Actual)

PRIMARY OUTCOMES:
exom | at day 0
  Exome measurement at the time of inclusion (D0) via a differential statistical analysis of the "burden" type aimed at comparing the organization of the mutational load between the two study groups

SECONDARY OUTCOMES:
exome variations | at day 0
  Identification of "Group1" specific candidate variant(s)/gene(s)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France, France

IPD SHARING:
Plan to Share IPD: No